A double-blind, randomized investigator-initiated study to determine the safety and the effect of Diamyd® in combination with Vitamin D on the progression to type 1 diabetes in children with multiple islet cell autoantibodies.

Study code: DiAPREV -IT 2

Phase IIa study

STATISTICAL ANALYSIS PLAN



| Signatures: | |
|-----------------------------------------------------|------|
| Statistical Analysis Plan was prepared by: | |
| Study Statistician<br>4Pharma Ltd | Date |
| Statistical Analysis Plan was reviewed/approved by: | |
| Senior Statistician<br>4Pharma Ltd | Date |
| CEO, Diamyd Medical AB | Date |
| Principal Investigator | Date |



# **Table of Contents**

| 1 A | Abbreviations | .4 |
|---|---|---|
| 2 S | Study objective(s)4 | |
| 3 D | Design and type of the study | .4 |
| 3.1 | Randomization and blinding | |
| 4 S | tudy variables | .5 |
| 5 S | ample size considerations | .5 |
| 6 S | tatistical hypotheses | .5 |
| 7 A | analysis sets | .6 |
| 7.1 | Intention to Treat Population (ITT) | |
| 7.2 | <b>→</b> 1 | |
| 7.3 | | |
| 7.4 | 7 1 | |
| | General statistical considerations | |
| | Demographic and other baseline characteristics | |
| 10 | Concomitant medication/treatment | |
| 11 | Extent of exposure and compliance | |
| 12 | Analysis of efficacy | |
| 12.<br>12. | | |
| 12 | | |
| 12 | | |
| 13 | Analysis of safety | |
| 13. | · | |
| 13. | | |
| 13. | , , , , | |
| 13.4 | 7 71 7 1 1 | |
| 13.:<br>13.: | <b>,</b> | |
| | · | |
| 14 | Completion and premature discontinuation | |
| 15 | Post diagnosis intervention and follow-up | |
| 16 | Deviations from the analyses planned in the study protocol | |
| 17 | Execution of statistical analyses | |
| 18 | Hardware and software | |
| 19 | References | |
| 20 | Appendices | |
| 20.<br>20. | | |
| ZU., | Z rapie and figure plan | 1 I |



#### 1 Abbreviations

AE Adverse Event

AUC Area Under the Curve

BDR Blind Data Review

DSMB Data Safety Monitoring Board

FPIR First-phase insulin response

HbA1c Hemoglobin A1c

ITT Intent to Treat

IvGTT Intravenous Glucose Tolerance Test

OGTT Oral Glucose Tolerance Test

PP Per-protocol

SAE Serious Adverse Event SAP Statistical Analysis Plan

#### 2 Study objective(s)

The purpose of the study is to assess the safety and efficacy of Diamyd $^{\otimes}$  20  $\mu g$  + vitamin D (2000 IU/day) in comparison with placebo + vitamin D (2000 IU/day) in non-diabetic children with multiple islet autoantibodies.

The primary objective of the study is to evaluate if Diamyd<sup>®</sup>, in children treated with relatively high doses of vitamin D, may delay or stop the autoimmune process leading to clinical type 1 diabetes in children with ongoing persistent beta cell autoimmunity as indicated by multiple positive islet cell autoantibodies.

The secondary objective is to demonstrate that Diamyd<sup>®</sup> is safe in children at risk for type 1 diabetes.

# 3 Design and type of the study

This is a phase IIa, double-blind, randomized, placebo-controlled, parallel group single centre study in children with multiple islet cell autoantibodies with a maximum of two-year follow-up.

### 3.1 Randomization and blinding

Eligible participants were randomized to active treatment or placebo, with 1:1 ratio. This randomization was stratified by glucose metabolism at baseline applying the following categorisation:

- A) Impaired glucose metabolism defined as low first phase insulin response on IvGTT ( $\leq$ 30) and/or an increased 30, 60, 90 min glucose values ( $\geq$  11.1 mmol/L) and/or 120 minutes glucose value ( $\geq$ 7.8 mmol/L) on OGTT, and/or HbA1c  $\geq$  39 and/or fasting glucose  $\geq$ 6.1 mmol/L
- B) Normal glucose metabolism



An independent statistician performed the randomization procedure. The randomization code for each child was preserved in envelopes in a locked safe. The treating physician had the possibility to break the code in cases of emergency. Further the Data Safety Monitoring Board (DSMB) had the possibility to request access to the randomization list.

### 4 Study variables

The following variables will be evaluated.

The demographic and baseline variables:

Age, Gender, Height, Weight, HLA genotypes, First degree relative or from general population, Autoantibodies, Other autoimmune diseases (celiac disease, thyroid disease).

The primary efficacy variable:

Type I diabetes status after 2-year follow-up

The secondary efficacy variables:

Proportion of children who progress from normal to impaired glucose metabolism and proportion of children who progress from impaired to more severely impaired glucose metabolism

The exploratory efficacy variables:

C-peptide, oGTT/IvGTT, plasma glucose, HbA1c

The safety variable:

Adverse events (AE), safety laboratory, physical and neurological examination, vital signs, GADA titers, isotype, epitope and affinity, anti-idiotypic antibodies, injection site reactions

#### 5 Sample size considerations

The planned sample size of the study was 80 children, 40 in each of the study arms. This sample size was based on the expectation that 50% of the untreated children with multiple autoantibodies will develop type 1 diabetes within 5 years. This frequency had previously been reported equal among relatives to diabetes patients and in the general population. If 20% of the treated children would develop type 1 diabetes within the same period of time, there would have been a power of 82% with alpha=5% with a group of 40+40=80 children. P value <0.05 was to be used as the significance level.

However, the study was stopped prematurely ending up with a total sample size of 29 children. The study was stopped due to negative results received from another similar study (DiAPREV/2008). In that study no effect on delaying or preventing type 1 diabetes with Diamyd®-treatment was shown, while GADA increased in the study patients. Since the cohort of children, inclusion and exclusion criteria and dose of Diamyd® were all equal in DiAPREV/2008 and DiAPREV-IT 2, it is not probable that the current study would show that Diamyd® would delay or prevent type 1 diabetes, but it may have effects on the immune system that can be explored in mechanistic studies.

#### 6 Statistical hypotheses

As the study was stopped prematurely with limited number of children within both treatment arms, no formal statistical hypotheses are defined.



# 7 Analysis sets

The database will be reviewed in a blinded manner prior to database lock. Patients are assigned to the respective analysis sets depending on the observed protocol violations.

## 7.1 Intention to Treat Population (ITT)

The ITT-population comprises all randomized (as planned) subjects.

# 7.2 Full Analysis Population

The Full Analysis Set (FAS) is a subset of ITT and comprises of all subjects who received any study drug and who participated in at least one post-baseline assessment. FAS is the primary efficacy population.

# 7.3 Per protocol (PP) Population

The PP population comprises of all subjects who did not substantially deviate from the protocol as to be determined on a per-subject basis. The PP population is used for sensitivity purposes.

# 7.4 Safety Population

The Safety Population comprises of all subjects who received at least one administration of the study drug at any dosage.

#### 8 General statistical considerations

Descriptive statistics include at least the number of participants, mean, standard deviation (SD), minimum, median and maximum for continuous variables, and frequencies and percentages for categorical variables. Line listings of all participants are provided as well.

Missing values will not be imputed in the analyses.

The table and figure plan is presented in Appendix 18.2.

# 9 Demographic and other baseline characteristics

All background and other baseline characteristics will be tabulated with descriptive statistics. Medical history will be summarized with frequency distributions including both event and subject counts. Tabulations will be conducted by treatment group. No statistical tests will be carried out for any baseline measures between the treatments.

#### 10 Concomitant medication/treatment

Concomitant medication and treatments will be summarized overall and by treatment group using ATC classification.



### 11 Extent of exposure and compliance

The extent of exposure and treatment compliance will be summarized descriptively overall and by treatment group.

#### 12 Analysis of efficacy

Descriptive statistics of all the efficacy data will be presented by visit and treatment group. ITT-population will serve as the primary efficacy population.

# 12.1 Primary efficacy variables

The primary efficacy variable is the type 1 diabetes status (with vs without type 1 diabetes) at the end of the two-year follow-up. The proportion of children developing clinical type 1 diabetes during the two-year follow-up will be summarized with frequency tables. The proportions of children with type 1 diabetes will also be summarized for other study visits by treatment group. The analysis will be conducted for both ITT and PP populations.

In addition, time to the development of type 1 diabetes up to 2 years will be graphically illustrated by Kaplan-Meier curves by treatment.

# 12.2 Secondary efficacy variables

The secondary efficacy variables are the proportion of children who have progression from normal to impaired glucose metabolism (within children with normal glucose metabolism at screening) and the proportion of children who have progression from already impaired glucose metabolism from one or several criteria to additional signs of reduced glucose metabolism (within children with impaired glucose metabolism at screening).

Impaired glucose metabolism is defined as acceptance of at least one of the following criterion; a) F-glucose  $\geq 6.1 \text{ mmol/L}$ , b) maximum p-glucose at 30, 60, 90 minutes  $\geq 11.1 \text{ mmol/L}$  in the OGTT, c) 120 min p-glucose  $\geq 7.8 \text{ mmol/L}$  on OGTT, d) HbA1c  $\geq 39 \text{ mmol/mol}$ .

Both the secondary efficacy variables will be summarized descriptively by visit and treatment group.

# 12.3 Subgroup analysis

Subgroup analysis will be conducted for the primary and secondary efficacy variables, so that the above-mentioned analyses will also be assessed by HLA genotype (DR3-DQ2, present/absent). The DR3-DQ2 subgroup will be derived from the database so that patients that have HLA-DQ haplotype of DQ2 (DQ2/8 or DQ2/x) are classified as DR3-DQ2 (present) and the ones without DQ2 (DQ2.2/8; DQ8/8 or DQ8/x) are classified as DR3-DQ2 (absent).



### 12.4 Exploratory efficacy variables

The exploratory efficacy variables include

- 1) first-phase insulin response (FPIR) and K-value from IvGTT
- 2) fasting, maximum, 2 hours and AUC<sub>0-120min</sub> C-peptide levels from OGTT,
- 3) fasting, maximum, 2 hours and AUC<sub>0-120min</sub> plasma-glucose from OGTT,
- 4) HbA1c (mmol/mol),
- 5) Fasting and AUC<sub>0-120min</sub> insulin levels from OGTT,
- 6) AUC<sub>90min</sub> of C-peptide, glucose and insulin from IvGTT

All the exploratory efficacy variables will be summarized descriptively including both the absolute and change from baseline values by visit and treatment group if feasible. In addition, the endpoints will be illustrated graphically if feasible.

The AUC values for C-peptide, plasma glucose and insulin will be calculated applying linear trapezoidal rule. In case of single missing time points for the C-peptide/plasma-glucose/insulin are detected, it will be assumed that missing values fall linearly between existing data points. In case the 0 min timepoint is missing, the corresponding AUC is set to missing.

# 13 Analysis of safety

All safety analyses will be conducted for the Safety population.

# 13.1 Adverse events

All adverse events (AEs) will be tabulated (according to the MedDRA dictionary) by treatment group, system organ class (SOC), preferred term (PT), severity and causality. Both participant and event counts will be calculated. For participants with more than one occurrence of the same preferred term, the strongest causality and severity will be used when participant counts are reported.

In addition, serious adverse events (SAE) and adverse events leading to discontinuation will be reported separately.

#### 13.2 Laboratory safety variables

Descriptive statistics of laboratory safety variables (hematology, chemistry and urine analyses) will be presented by visit and treatment group, together with the changes from baseline (pre-dose) values.

# 13.3 Physical and neurological examination, vital signs

Vital signs (blood pressure, heart rate) will be summarized descriptively by visit and treatment group, together with changes from baseline (pre-dose). The abnormal findings in physical and neurological examinations will be presented as frequencies and percentages by visit and treatment group.



### 13.4 GADA titers, isotype, epitope and affinity, anti-idiotypic antibodies

GADA titers, isotype, epitope and affinity, anti-idiotypic antibodies (GADA (U), IA-2A (U), IAA ny (U/mL), ZnT8ArgA (U), ZnT8TrpA (U), ZnT8GluA (U)) will be summarized descriptively by visit and treatment group. In addition, GADA titers will be illustrated graphically.

#### 13.5 Autoimmunity other than diabetes

Autoantibodies to Thyroid peroxidase (TPO), Thyroglobulin (Thgl) and Tissue transglutaminase (tTg), (Thyroid peroxidase Ab (U), Thyroglobulin Ab (U), tTG IgA (U) and tTG IgG (U) together with TSH (mU/L) and Free T4 (pmol/L), will be summarized descriptively at visit 0, 12 months and 24 months by treatment group.

### 13.6 Injection site reactions

The number of injection site reaction by severity will be summarized by visit and treatment group.

### 14 Completion and premature discontinuation

Completion and premature discontinuation will be listed. The reasons for premature discontinuation will be presented.

#### 15 Post diagnosis intervention and follow-up

Study participants who developed type 1 diabetes during the study period were offered to participate in a post diagnosis intervention and follow up protocol. The collected post diagnosis data from the included participants will be summarized using data listings.

#### 16 Deviations from the analyses planned in the study protocol

Due to the premature stop of the study, all the formal statistical analyses were removed from the statistical analysis plan compared to the protocol.

#### 17 Execution of statistical analyses

Statistical analyses will be performed by 4Pharma Ltd.

#### 18 Hardware and software

Statistical analysis, tables and patient data listings will be performed with SAS® version 9.4 for Windows (SAS Institute Inc., Cary, NC, USA). Pharmacokinetic parameters (AUC<sub>0-120min</sub> for C-peptide, glucose and insulin) will be calculated using Phoenix WinNonlin software (version 8.1; Certara USA, Inc; Princeton; NJ; USA).

#### 19 References

Clinical Study Protocol, Version 3 (28.08.2017)

#### 20 Appendices



# 20.1 Schedule of assessments

| Event | Visit 0<br>Information<br>and consent | Visit 1 Day 1 30 +/- 7 days from visit 0 | Visit 2<br>Month 1<br>30 +/-7 days<br>from visit 1 | Visit 3 Month 3 3 months +/- 14 days from visit 1 | Visit 4 Month 6 6 months +/- 14 days from visit 1 | Visit 5 Month<br>9<br>9 months<br>+/- 14 days<br>from visit 1 | Visit 6<br>Month 12<br>12 months<br>+/- 14 days<br>from visit 1 | 5 Years Follow up<br>Every 3rd or 6th month<br>Every visit<br>+/- 14 days<br>from visit 1 |
|---|---|---|---|---|---|---|---|---|
| Informed Consent | X | | | | | | | |
| Randomization | | X | | | | | | |
| Diamyd/Placebo<br>Administration | | X | X | | | | | |
| Start of Vitamin D | X | | | | | | | |
| Medical History | X | | | | | | | |
| General Physical Exam | X | X | X | X | X | | X | Last visit |
| Concomitant Medication | X | X | X | X | X | | X | Every 6th month |
| Weight, Height | X | X | X | X | X | | X | Every 6th month |
| Vital signs (BP) | X | X | X | X | X | | X | Every 6th month |
| Blood Sampling: | | | | | | | | |
| Hematology, chemistry, including calcium | X | X | X | X | X | X | X | Every 3rd month |
| 25 OH-vitamin D3 | X | X | | | X | | X | Every 6th month |
| Cellular analyses | X | | X | | X | | X | Every 6th month |
| GADA, IA-2A, ZnT8A,<br>IAA | X | X | X | X | X | X | X | Every 3rd month |
| C-peptide | X<br>Fasting +<br>stimulated | X<br>Fasting +<br>stimulated | X<br>Random | X<br>Random | X<br>Fasting +<br>stimulated | X<br>Random | X<br>Fasting +<br>stimulated | Every 6th month Fasting + stimulated |
| HbA1c | X | X | X. | X | X | X | X | Every 3rd month |
| Plasma Glucose | X | X | X | X | X | X | X | Every 3rd month |
| OGTT/IvGTT | IvGTT | OGTT | | | OGTT | | IvGTT | Every 6th month IvGTT/OGTT |
| TPOAb, ThglAb, tTGAb | X | | | | | | X | Every 12th month |
| Urine Analysis | X | X | X | X | X | | X | Every 6th month |
| Neurological Assessment | X | | X | X | X | | X | Last visit |
| Injection Site Inspection | | X | X | X | X | | | |
| Adverse Events | | X | X | X | X | | X | Last visit |
| Diary | | X | X | X | X | | X | Last visit |
| Questionnaire to child about the study procedures | | X | | | | | | Last visit |

**Sponsor:** Diamyd Medical AB Final 5.5.2020 **Study:** DiAPREV-IT 2



| 20.2 Table and figure plan | |
|---|---|
| 14.1 | Demographic and Baseline Characteristics |
| Table 14.1.1 | Disposition of patients (Total population) |
| Table 14.1.2 | Analysis sets (Total population) |
| Table 14.1.3 | Descriptive statistics of demographic variables (ITT) |
| Table 14.1.4 | Medical history (ITT) |
| Table 14.1.5 | Current medical conditions at baseline (ITT) |
| Table 14.1.6 | Concomitant medication (ITT) |
| 14.2 | Efficacy |
| 14.2.1 | Primary efficacy analyses |
| Table 14.2.1.1 | Type 1 diabetes status by treatment and visit (ITT) |
| Table 14.2.1.2 | Type 1 diabetes status by treatment and visit within subgroup (ITT) |
| Table 14.2.1.3 | Time to development of type 1 diabetes (ITT) |
| Table 14.2.1.4 | Time to development of type 1 diabetes by subgroup (ITT) |
| 14.2.2 | Secondary efficacy analyses |
| Table 14.2.2.1 | Number of children developing impaired glucose metabolism (ITT) |
| Table 14.2.2.2 | Number of children developing impaired glucose metabolism by subgroup (ITT) |
| Table 14.2.2.3 | Number of children having progressive impaired glucose metabolism (ITT) |
| Table 14.2.2.4 | Number of children having progressive impaired glucose metabolism by subgroup (ITT) |
| 14.2.3 | Exploratory efficacy analyses |
| Table 14.2.3.1 | Descriptive statistics of first-phase insulin response (FPIR) and K-value from IvGTT by treatment and visit (ITT) |
| Table 14.2.3.2 | Change from baseline in first-phase insulin response (FPIR) and K-value from IvGTT by treatment and visit (ITT) |
| Table 14.2.3.3 | C-peptide concentrations from OGTT by treatment, visit and timepoint (ITT) |
| Table 14.2.3.4 | Maximum and AUC0-120min C-peptide values from OGTT by treatment and visit (ITT) |
| Table 14.2.3.5 | Change from baseline in fasting, maximum and 2 hours C-peptide (OGTT) by treatment, visit and timepoint (ITT) |
| Table 14.2.3.6 | P-glucose concentrations from OGTT by treatment, visit and timepoint (ITT) |
| Table 14.2.3.7 | Maximum and AUC0-120min P-glucose values from OGTT by treatment and visit (ITT) |
| Table 14.2.3.8 | Change from baseline in fasting, maximum and 2 hours P-glucose (OGTT) by treatment, visit and timepoint (ITT) |
| Table 14.2.3.9 | HbA1c concentrations by treatment, visit and timepoint (ITT) |
| Table 14.2.3.10 | Change from baseline in HbA1c concentration by treatment, visit and timepoint (ITT) |
| Table 14.2.3.11 | Insulin concentrations from OGTT by treatment, visit and timepoint (ITT) |
| Table 14.2.3.12 | Maximum and AUC0-120min Insulin values from OGTT by treatment and visit (ITT) |
| Table 14.2.3.13 | Change from baseline in fasting and maximum Insulin concentration (OGTT) by treatment, visit and timepoint (ITT) |
| Table 14.2.3.14 | C-peptide concentrations from IvGTT by treatment, visit and timepoint (ITT) |
| Table 14.2.3.15 | AUC0-90min C-peptide values from IvGTT by treatment and visit (ITT) |
| Table 14.2.3.16 | Glucose concentrations from IvGTT by treatment, visit and timepoint (ITT) |
| Table 14.2.3.17 | AUC0-90min Glucose values from IvGTT by treatment and visit (ITT) |
| Table 14.2.3.18 | Insulin concentrations from IvGTT by treatment, visit and timepoint (ITT) |
| Table 14.2.3.19 | AUC0-90min Insulin values from IvGTT by treatment and visit (ITT) |



| 14.3 | Safety |
|---|---|
| 14.3.1 | Adverse events |
| Table 14.3.1.1 | Summary of adverse events (Safety) |
| Table 14.3.1.2 | Adverse events by SOC and PT (Safety) |
| Table 14.3.1.3 | Adverse events by SOC, PT and severity (Safety) |
| Table 14.3.1.4 | Adverse events by SOC, PT and causality (Safety) |
| Table 14.3.1.5 | Serious adverse events (Safety) |
| Table 14.3.1.6 | Adverse events leading to discontinuation (Safety) |
| 14.3.2 | Laboratory safety variables |
| Table 14.3.2.1 | Summary of safety laboratory - Hematology (Safety) |
| Table 14.3.2.2 | Summary of safety laboratory - Clinical chemistry (Safety) |
| Table 14.3.2.3 | Summary of safety laboratory - Urinanalysis (Safety) |
| 14.3.3 | Physical and neurological examination, vital signs |
| Table 14.3.3.1 | Physical examination by treatment and visit (Safety) |
| Table 14.3.3.2 | Neurological examination by treatment and visit (Safety) |
| Table 14.3.3.3 | Vital signs (blood pressure, heart rate) by treatment and visit (Safety) |
| Table 14.3.3.4 | Change from baseline in Vital signs (blood pressure, heart rate) by treatment and visit (Safety) |
| 14.3.4 | GADA titers, isotype, epitope and affinity, anti-idiotypic antibodies |
| Table 14.3.4.1 | Descriptive statistics of GADA (U) by treatment and visit |
| Table 14.3.4.2 | Descriptive statistics of IA-2A (U), IAA ny (U/mL) by treatment and visit |
| Table 14.3.4.3 | Descriptive statistics of ZnT8ArgA (U), ZnT8TrpA (U), ZnT8GluA (U) by treatment and visit |
| 14.3.5 | Autoimmunity other than diabetes |
| Table 14.3.5.1 | Descriptive statistics of autoimmunity related autoantibodies by treatment and visit |
| 14.3.6 | Injection Site Reactions (Safety) |
| Table 14.3.6.1 | Injection site reactions (erythmea, oedema, haematoma, tenderness, pain, itching), pre-injection by visit and treatment (Safety) |
| Table 14.3.6.2 | Injection site reactions (erythmea, oedema, haematoma, tenderness, pain, itching), post-injection by visit and treatment (Safety) |
| 14.3.7 | Questionnaire to child about study procedures |
| Table 14.3.7.1 | Frequency table of child's assessment of study procedures (Safety) |
| 14.2 | Figures |
| Figure 14.2.1 | Kaplan-Meier curves of time to development of type 1 diabetes (ITT) |
| Figure 14.2.2 | C-peptide concentrations (OGTT - ITT) |
| Figure 14.2.3 | P-Glucose concentrations (OGTT - ITT) |
| Figure 14.2.4 | Insulin concentrations (OGTT - ITT) |
| Figure 14.2.5 | C-peptide concentrations (IvGTT - ITT) |
| Figure 14.2.6 | Glucose concentrations (IvGTT - ITT) |
| Figure 14.2.7 | Insulin concentrations (IvGTT - ITT) |
| Figure 14.2.8 | HbA1c concentrations (ITT) |



| 16.2 | Patient Data Listings |
|-------------------|-------------------------------------------------|
| Listing 16.2.1 | Protocol Deviations |
| Listing 16.2.2 | Demographic data |
| Listing 16.2.3 | Medical history |
| Listing 16.2.4 | Concomitant medications |
| 16.2.5 | Individual Efficacy Response data |
| Listing 16.2.5.2 | Glucose data (OGTT, IvGTT) |
| Listing 16.2.5.3 | C-peptide data (OGTT, IvGTT) |
| Listing 16.2.5.4 | Insulin data (OGTT, IvGTT) |
| Listing 16.2.5.5 | HbA1c data |
| Listing 16.2.6 | Adverse events |
| Listing 16.2.7 | Individual laboratory measurements by patient |
| Listing 16.2.8 | Physical, neurological examination, vital signs |
| Listing 16.2.9 | Injection site reactions |
| Listing 16.2.10 | Other safety variables |
| 16.2.11 | Post diagnosis data |
| Listing 16.2.11.1 | C-peptide, glucose, HbA1c |
| Listing 16.2.11.2 | MMTT-data |
| Listing 16.2.11.3 | Safety laboratory |
| Listing 16.2.11.4 | Physical, neurological examination, vital signs |
| Listing 16.2.11.5 | Adverse events |